CLINICAL TRIAL: NCT00566735
Title: The Use of Galantamine HBr (Reminyl) in Electroconvulsive Therapy: Impact on Mood and Cognitive Functioning
Acronym: Galantamine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Ortho-McNeil Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Principal Investigator, John D. Matthews, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2004-P-001051; GAL-EMR-4005 (Other: Janssen Pharmaceuticals)
Record Dates: First submitted 2007-12-03; First posted 2007-12-04 (Estimated); Results first posted 2012-12-03 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Major Depression; Bipolar Depression; Schizoaffective Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder; Psychotic Disorders | interventions — Galantamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- 2, Galantamine (Active Comparator)
  Interventions: Drug: Razadyne

INTERVENTIONS:
Drug: Razadyne — The starting dose of study medication is 4 mg twice a day
  Other Names: Galantamine
  Arms: 2, Galantamine
Drug: Placebo — 4 mg, 2 times a day
  Arms: 1

SUMMARY:
The purpose of the study is to see if galantamine HBr (Razadyne) is safe and can help treat problems with thinking and memory caused by electroconvulsive therapy (ECT).

ELIGIBILITY:
Inclusion Criteria:

* Criteria to enter the study include males and females between the ages of 18-90 (females must be post menopausal) and a DSM-IV diagnosis of Major Depressive Disorder, Major Depressive Disorder with psychotic features, Bipolar Disorder, depressed type, or Schizoaffective Disorder, depressed type (19).

Exclusion Criteria:

* DSM-IV diagnoses of dementia and its subtypes
* Substance use disorder (active use within the last 6 months)
* Organic mental disorders; seizure disorder
* Unstable physical disorder or physical disorder judged to significantly affect the central nervous system function
* A heart rate of <60
* A systolic blood pressure < 90
* Heart block
* Pre-existing sick-sinus
* Chronic treatment with beta blockers
* Any cardiac arrythmia
* Hypotension
* Coronary artery disease
* Liver and renal function impairment
* Urge incontinence, colitis Crohn's disease, GI motility disorders, asthma and COPD
* Treatment with anti-cholinergic and cholinomimetic medications; and
* Female patients who are pregnant.
* Additionally, women subjects must be postmenopausal, surgically sterile, or using prescription oral contraceptives (e.g. estrogen-progestin combinations) , contraceptive implants (e.g. NorplantTM, DepoProveraTM ), or transdermally delivered contraceptives (Ortho EvraTM) before entry and throughout the study; and have a negative serum b-HCG pregnancy test at screening.

Note: Abstinence and the use of double barrier contraceptive methods are not acceptable in this study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2004-07; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D Matthews, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Patients with major depression, bipolar disorder (depressed type) or schizoaffective disorder (depressed type) received placebo (sugar pills) and treatment-as-usual electroconvulsive therapy.
- Galantamine: Patients with major depression, bipolar disorder (depressed type) or schizoaffective disorder (depressed type) received galantamine tablets 4 milligrams twice daily (increased every three days until a target of 8 milligrams twice daily) and treatment-as-usual electroconvulsive therapy.
Period: Overall Study
Arm/Group | Placebo | Galantamine
Started | 20 | 19
Withdrew Before Baseline Measures | 2 | 7
Completed | 18 (2 participants withdrew before baselines. Therefore, 18 participants will be included in baselines.) | 12 (7 participants withdrew before baselines. Therefore, 12 participants will be included in baselines.)
Not Completed | 2 | 7
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Refused neuropsychological testing | 2 | 5
Not completed — Switched into a manic episode | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Galantamine | Total
Number analyzed (Participants) | 18 | 12 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 9 | 23
  >=65 years | 4 | 3 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 6 | 17
  Male | 7 | 6 | 13
Wechsler Abbreviated Scale of Intelligence (WASI) [Mean (Standard Deviation); unit: WASI Score] — The WASI is a standardized measurement of intelligence quotient (IQ). Scores range from 1 to 160, with 100 signifying average intelligence, scores above 140 signifying superior intelligence, and scores below 40 signifying severe intellectual impairment.
  WASI Score | 102.16 (18.21) | 104.57 (12.35) | 103.12 (15.87)
Hamilton Depression Rating Scale 17 (HAM-D-17) [Mean (Standard Deviation); unit: HAM-D-17 Score] — This scale is a rater-administered assessment of depression severity and improvement. Scores range from 0 (not depressed) to 52 (severely depressed).
  HAM-D-17 Score | 27.33 (4.33) | 24.53 (4.33) | 26.21 (4.33)
Subjective Mood [Mean (Standard Deviation); unit: Subjective Mood Score] | 8.0 (1.54) | 7.88 (1.93) | 7.95 (1.70)
Clinical-Global Impressions - Severity (CGI-S) [Mean (Standard Deviation); unit: CGI-S Score] — This scale is a rater-administered assessment of severity of symptoms. 1 = Normal, not ill at all; 2 = Borderline ill; 3 = Mildly ill; 4 = Moderately ill; 5 = Markedly ill; 6 = Severely ill; 7 = Among the most extremely ill patients
  CGI-S Score | 4.75 (0.62) | 4.41 (0.87) | 4.61 (.72)
Modified Mini Mental Status Exam (3MSE) [Mean (Standard Deviation); unit: 3MSE Score] — The 3MSE is a rater-administered test that assesses a broad variety of cognitive functioning. Scores range from 0 to 30. Scores greater than 25 indicate a normal cognition. Below this, scores can indicate severe (≤9 points), moderate (10-20 points) or mild (21-24 points) cognitive impairment.
  3MSE Score | 91.72 (8.05) | 90.41 (5.48) | 91.20 (7.02)

OUTCOME MEASURES:

1. Primary Outcome: Number of Side Effects
Description: This measure refers to the number of reported side effects experienced by participants during the study. The side effects were nausea, headache, dizziness, diarrhea, and vomiting.
Time Frame: Participants were followed for the duration of hospital stay, an average of 3 weeks
Measure: Number; unit: Number of reported side effects
Arm/Group | Placebo | Galantamine
Number analyzed (Participants) | 18 | 12
Number of reported side effects | 19 | 13

2. Secondary Outcome: Cognitive Functioning
Description: This measure refers to participants' scores on the Delayed Memory Index (DMI) compared from baseline (before first ECT) to discharge (after last ECT). The score can range from 40 to 137. The higher the score, the better, in terms of cognitive functioning.
Time Frame: Participants were questioned at baseline and after their last electroconvulsive therapy treatment
Measure: Mean (Standard Deviation); unit: Score on the DMI
Arm/Group | Placebo | Galantamine
Number analyzed (Participants) | 18 | 12
Score on the DMI
  Pre-ECT | 80.33 (17.87) | 88.75 (15.64)
  Post-ECT | 68.50 (22.65) | 88.17 (19.84)
Statistical Analysis 1: Comparison: Placebo vs Galantamine; Independent t-test to assess differences between the placebo and galantamine groups in regard to pre- and post-ECT scores on the Delayed Memory Index (DMI); Test type: Superiority or Other; p < 0.05, t-test, 1 sided; Degrees of freedom = 28

3. Secondary Outcome: Baseline Depressive Symptoms
Description: This measure refers to the Hamilton Rating Scale for Depression-17 scores (HAM-D-17) which can range from 0 to 50, with <7 referring to mild-to-no depression, and >23 referring to severe depression.
Time Frame: Participants were questioned at baseline
Measure: Mean (Standard Deviation); unit: Score on the HAM-D-17
Arm/Group | Placebo | Galantamine
Number analyzed (Participants) | 18 | 12
Score on the HAM-D-17 | 24.53 (4.33) | 27.33 (4.33)

ADVERSE EVENTS:
Arm/Group | Placebo | Galantamine
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 19/19 | 13/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=19) | Galantamine (N=18)
nausea (General disorders) | 3 (3) | 2 (2)
headache (General disorders) | 5 (5) | 3 (3)
dizziness (General disorders) | 4 (4) | 3 (3)
diarrhea (Gastrointestinal disorders) | 4 (4) | 2 (2)
vomiting (Gastrointestinal disorders) | 3 (3) | 3 (3)

LIMITATIONS AND CAVEATS:
The limitations of this study include a small sample size, absence of an optimal galantamine dose determination, and the inclusion of a heterogenous population including MDD, bipolar disorder, and schizoaffective order.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No